CLINICAL TRIAL: NCT02937779
Title: Tenofovir As Prevention Of Hepatitis b Mother-to-child Transmission
Acronym: TA-PROHM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 12345
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Hepatitis B Chronic Infection; Pregnancy
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBs Ag positive (Experimental): tenofovir disoproxil fumarate 300 mg one tablet once daily from 24 weeks of amennorrhea to 6 weeks post-partum for positive Hbe Ag women.
  No treatment for negative HBe Ag women
  Interventions: Drug: Tenofovir disoproxil fumarate; Device: Rapid tests HBe Ag

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — tenofovir disoproxil fumarate 300 mg one tablet once daily from 24 weeks of amennorrhea to 6 weeks post-partum for HBe Ag positive women only.
  Other Names: TDF
Device: Rapid tests HBe Ag — For all HBs Ag positive women

SUMMARY:
The World Health Organization recommends that all high endemic countries for HBV infection based their mother to child transmission prevention strategies on vaccination of all children and administration of immunoglobulins (HBIG) to infants born to infected mothers in the first 24 hours after birth. Lack of access to antenatal screening and to HBIG significantly results in failure of this strategy in many countries. Moreover, despite sero-vaccination, 10 to 15% of infants of mothers that are positive for HBsAg and HBeAg are still infected, as high levels of HBV replication occurring in the third quarter of pregnancy act as a major risk factor.

The objective of this study is to assess the effectiveness of an operational strategy to prevent HBV mother-to-child transmission (MTCT) in Cambodia based on the use of rapid tests HBs Ag and HBe Ag to screen HBV infection and a treatment by TDF for patients with a positive HBeAg test with a "test and treat" strategy for those seen for Antenatal Care (ANC) from 24 weeks of amenorrhea. In all cases, vaccination of the newborn will be carried out according to the national protocol in Cambodia i.e. 4 injections at 24 hours, 6, 10 and 14 weeks of age.

A phase IV multicenter observational and interventional non randomized prospective study will be conducted in 4 maternity in Cambodia.

The primary outcome will be the proportion of active HBV infection in new-born at 6 months of life estimated by HBs Ag positivity.

The study will aim to document the acceptability and the operational implementation of the study using rapid tests usable in all health centers and a drug available in all the country thanks to HIV national program. The results will be helpful for Cambodian government in order to implement guidelines and algorithm follow-up for HBV-infected pregnant women.

DETAILED DESCRIPTION:
Principal objective: Assess the effectiveness of a strategy to prevent HBV mother-to-child transmission (MTCT) in Cambodia based on the use of rapid tests HBs Ag and HBe Ag to screen HBV infection and a treatment by TDF for patients with a positive HBeAg test with a "test and treat" strategy for those seen for Antenatal Care (ANC) from 24 weeks of amenorrhea.

Secondary objectives Assess the feasibility and acceptability for patients and health care providers of the rapid tests screening strategy Assess the acceptability of the test and treat strategy for patients seen after 24 weeks of amenorrhea Describe the HBV viral load (VL) decrease caused by the TDF Estimate the rate of HBV transmission to newborns according to the time spent on TDF as well as initial viral load level and delivery viral load level Estimate the rate of HBV transmission to newborns for HBe Ag negative women Describe the correlation between HBV viral load level and HBe Ag status Describe subgroups of mothers and new-borns for which the strategy seems more effective Assess TDF safety in mothers Analyse the cost-effectiveness of the strategy compare to international guidelines (WHO, APASL)

Each woman will be informed of the objectives and the total duration of the study as well as the benefits and risks to participate. An information sheet in Khmer will be given to each woman. The study will be composed of two phases of information's and consent. The first one will be done during the HBs Ag screening using rapid test; the screening will be proposed to all pregnant women attending ANC in one of the affiliated centres. The second phase will be done during the inclusion visit and will concern only HBs Ag positive women. The study will concern only HBs Ag positive women with 1) follow up of all HBsAg positive women from inclusion up to 6 months postpartum 2) For HBeAg positive women, initiation of treatment by fumarate de tenofovir disoproxil (Viread®), with a daily administration of one 300mg pill. Women will be treated from 24 weeks of amenorrhea until 6 weeks post-partum. For women with first ANC after 24 weeks of amenorrhea, treatment will begin the day of inclusion. Treatment will be given for 4 weeks and adherence will be estimated. In all cases, vaccination of the newborn will be carried out according to the national protocol in Cambodia i.e. 4 injections at 24 hours, 6, 10 and 14 weeks of age.

A total of 933 positive HBs Ag pregnant women will be enrolled including 280 HBe Ag positive women and 653 HBe negative women.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old the day of inclusion
* Pregnancy
* Positive HBs Ag
* Informed consent obtained with information sheet given and explained and the consent form signed by the participant of the project investigator at the latest the day of the inclusion

Exclusion Criteria:

* Women refusing HBs Ag test
* HIV co-infection
* HCV co-infection
* HBV treatment ongoing at the day of inclusion
* Creatinine clearance < 30 mL/min
* Severe gravidic disease present at inclusion involving life threatening to the mother and/or the child
* Evidence of pre-existing fetal anomalies incompatible with the child's life
* Imminent child's birth defined as cervix dilatation up to 7 centimeters
* Intention to deliver in a maternity not linked to the study
* Any concomitant medical condition that, according to the clinical site investigator would contraindicate participation in the study.
* Concurrent participation in any other clinical trial without written agreement of the two study teams

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 933 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of active HBV infection in new-born at 6 months of life | 6 months post-partum
  The proportion will be estimated by HBs Ag positivity

SECONDARY OUTCOMES:
Process and acceptability of the screening phase | Enrollement
  Proportion of women with screening proposed among those eligible in antenatal consultation (ANC)
Process and acceptability of the screening phase | Enrollement
  Proportion of women with a done screening among those to whom screening was proposed
Process and acceptability of the screening phase | Enrollement
  Proportion of women with a given results in less than one day among those to whom the test was made
Process and acceptability of the screening phase | Enrollement
  Care-giver satisfaction regarding the strategy (estimated by questionnaires)

OTHER OUTCOMES:
Process and acceptability of the drug's intervention | Enrollement
Proportion of women with viral load > 6 Log among those HBe Ag negative | Enrollement
Proportion of new-born with positive HBs Ag at 6 months according to treatment duration, initial and delivery viral load level | 6 months post-partum
Decrease curve of HBV VL after TDF initiation over time | From enrollement to 8 weeks or 6 months post-partum
Occurrence of maternal adverse events including serious adverse events and adverse events grade 3 or 4 | From enrollement to 6 months post-partum
Proportion of women needing treatment continuation in post-partum among those to whom treatment was initiated | 6 weeks post-partum
Occurrence of acute exacerbation after treatment interruption | From 8 weeks post-partum to 6 months post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Samsorphea CHHUN, MD, Principal Investigator — Calmette Hospital
Locations (3):
- Cambodia (3):
  - Kampong Cham Provincial Hospital, Kampong Cham
  - Calmette Hospital, Phnom Penh
  - National Mother and Child Health Center, Phnom Penh

REFERENCES:
- [Derived] Segeral O, Dim B, Durier C, Nhoueng S, Chhim K, Sovann S, Yom S, Vong C, Yin S, Ros B, Ky V, Pech S, Nem B, Hout K, Guillebaud J, Ear E, Caroupaye-Caroupin L, Rekacewicz C, Fernandez L, Laurent D, Yay C, Kim R, Meyer L, Chhun S; Laurence Borand for the ANRS-MIE TA PROHM Study Group. Immunoglobulin-free strategy to prevent HBV mother-to-child transmission in Cambodia (TA-PROHM): a single-arm, multicentre, phase 4 trial. Lancet Infect Dis. 2022 Aug;22(8):1181-1190. doi: 10.1016/S1473-3099(22)00206-7. Epub 2022 May 25. PMID 35643089